CLINICAL TRIAL: NCT05256329
Title: A Predictive Score for Arterial Thrombosis Associated With Cancer. The Prospective COMPASS- Arterial Cancer Associated Thrombosis Study
Brief Title: A Predictive Score for Arterial Thrombosis Associated With Cancer
Acronym: COMPASS-ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Institut Universitaire de Cancérologie, Sorbonne University (Unknown); Third Department of Medicine, Sotiria General Hospital (Unknown); Oncology Department, Hippokration Hospital (Unknown); Metaxa Hospital, Cardiology Department, Greece (Unknown)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Professor of Cardiology, National and Kapodistrian University of Athens
Other Study IDs: 14281
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncology patients: Patients suffering from specific solid cancers or hematological malignancies

SUMMARY:
Cancer is associated with an increased incidence of thrombosis and thromboembolic events are one of the leading causes of morbidity and mortality in this population. The main consideration has been given to venous thromboembolic events (VTEs); arterial thrombotic events (ATEs) have more recently been recognized to precede cancer diagnosis and/or follow it as a serious complication. Thus, while plausible, the relationship between cancer and arterial thrombosis is less well established than for VTE. We sought to undertake the COMPASS-ARTeCAT (Comparison of Methods for thromboembolic risk assessment with clinical Perceptions and AwareneSS in real life patients- Arterial Cancer Associated Thrombosis) study aiming to identify the most clinically relevant clinical predictors of arterial thrombosis in ambulatory patients with specific types of cancer who are going to start or have already started anticancer treatment. This study aims to evaluate the incidence and the association between arterial thromboembolism and occult cancer. Moreover, this study will provide a risk assessment model (RAM) for arterial thrombosis applicable to cancer patients at any time after anticancer therapy initiation

DETAILED DESCRIPTION:
Cancer is associated with an increased incidence of thrombosis and thromboembolic events are one of the leading causes of morbidity and mortality in this population. The main consideration has been given to venous thromboembolic events (VTEs); arterial thrombotic events (ATEs) have more recently been recognized to precede cancer diagnosis and/or follow it as a serious complication. Thus, while plausible, the relationship between cancer and arterial thrombosis is less well established than for VTE.

The heightened risk for VTEs in outpatients who receive anticancer treatment has been extensively investigated and associated to the histological type of the malignancies, the stage of the disease, the time since cancer diagnosis and the expanding armamentarium of chemotherapeutic agents. Patients' intrinsic risk factors and particularly, the presence of cardiovascular risk factors and personal history of VTE, as well as other underlying comorbidities (i.e. recent hospitalization for acute medical illness, acquired or hereditary thrombophilia, autoimmune disease) are determinant clinical predictors for VTE and have been included to the most recent risk assessment models (RAMs) for patients with common solid tumors (i.e. breast, lung, ovarian or colon cancers) or hematological malignancies (i.e. lymphoma). In specific, the COMPASS-CAT (Comparison of Methods for thromboembolic risk assessment with clinical Perceptions and AwareneSS in real life patients-Cancer Associated Thrombosis) and ThroLy (Thrombosis Lymphoma) scores are derived from prospective multicentric observational studies specifically designed to evaluate the clinical relevance of predictors related to cancer characteristics, patients' intrinsic risk factors and anticancer treatment related risk factors. The COMPASS-CAT score for VTE is applicable to cancer patients at any time after anticancer therapy initiation providing a global evaluation of VTE risk, feasible in real life conditions of medical oncology practice. This score been externally validated in about 4000 patients and showed similar accuracy, sensitivity and specificity as compared to the ones reported in the initial derivation study. Thus, the methodological design applied in the COMPASS-CAT study (prospective multicenter observational study with symptomatic and documented end point of thrombosis and elaboration of an extensive CRF including all known cancer related and patient- related risk factors for thrombosis) leads to an accurate RAM.

Taking into consideration that clinical research in the field of risk assessment tools in cancer associated arterial thrombosis is delayed compared to the respective in cancer associated VTE, we sought to undertake the COMPASS-ARTeCAT (Comparison of Methods for thromboembolic risk assessment with clinical Perceptions and AwareneSS in real life patients- Arterial Cancer Associated Thrombosis) study aiming to identify the most clinically relevant clinical predictors of arterial thrombosis in ambulatory patients with specific types of cancer who are going to start or have already started anticancer treatment. The COMPASS-ARTeCAT study will be a multicenter, prospective, longitudinal, non-interventional study undertaken in patients suffering from specific solid cancers or hematological malignancies and will derive to a new RAM for identification of patients at risk for arterial thrombosis which will be applicable during patients' journey in the oncological context.

Materials and methods Study Design and Participants. This study is an investigator-initiated multinational, prospective, and non-interventional trial. Ambulatory cancer patients, with histologically confirmed solid cancer (breast, lung, gastric, colorectal, pancreatic, ovarian, prostate, or bladder cancer) or specific hematologic malignancy (Hodgkin and non-Hodgkin lymphoma or multiple myeloma), will be recruited and followed from January 2021 to January 2023. Patients diagnosed with multiple primary cancers during the study period will be assigned to the cancer type diagnosed first. The specific site definitions for cancer cohorts will be based on the International Classification of Diseases (ICD) for Oncology, third edition, site recode classification to identify the cancer population. Consecutive patients from the ambulatory anticancer clinics will be assessed for eligibility. Patients with: (a) age younger than 18 years, (b) life expectancy less than 3 months, (c) ongoing pregnancy, (d) recent (≤3 months) arterial thromboembolism and/or (e) major psychiatric disorder will be excluded from the study.

Patients at assessment for eligibility in the study will be receiving or will be scheduled to receive the recommended anticancer treatments according to the institutional practices. At the follow-up visits, at 3, 6, 12 and 24 months after inclusion, patients will be interviewed and clinical records will be analyzed regarding the occurrence of symptomatic arterial thrombosis, bleeding episodes, disease evolution, and anticancer treatments. During the study, investigators will be free to decide for antiplatelet and/or anticoagulation therapy according to local clinical practice and individual perception of the thrombotic risk. All patients enrolled in the study will provide written informed consent. The study protocol will be approved by the institutional review boards or ethics committees of all participating institutions.

Outcomes. The primary outcome of the study is a composite of symptomatic arterial thromboembolism, defined as any inpatient diagnosis of: 1) acute coronary syndrome (ACS) including ST- elevation myocardial infarction (STEMI), non-ST elevation MI (NSTEMI) or unstable angina (UA), 2) transient ischemic attack (TIA) or ischemic stroke or 3) other arterial thromboembolism (systemic embolism or mesenteric ischemia) defined according to the respective diagnostic criteria and recommendations. The secondary outcomes are peripheral arterial disease (diagnosis or progression) and hypertension (new or worsening).

Definitions for Key Predictors for arterial thrombosis. Eligible patients will be interviewed at the inclusion visit using a standardized clinical research form (CRF) with previously validated factors for arterial thromboembolism. The CRF will also assess the status of the oncological disease, the ongoing treatments and the values of common and routinely performed hemogram and laboratory parameters of liver and renal function measured within 1 week prior to enrollment. The body mass index (BMI) at the day of the assessment will be stratified into three groups: normal weight (BMI less than 25), overweight (BMI greater than or equal to 25 and less than 30), or obese (BMI greater than or equal to 30). The predictors "smoking", "hyperlipidemia," "hypertension", "diabetes mellitus", "family history of coronary artery disease (CAD)", as well as a background of "stroke," "CAD" and/or "peripheral artery disease (PAD)" will appear individually in the CRF, assessed at the inclusion point, and refer to objectively diagnosed conditions according to the respective diagnostic criteria. Separate variables will be created according to the number of risk factors coexisting in a patient (one, two, three, or four risk factors together) and their relative risk for arterial thrombosis will be evaluated in the multivariate analysis. The "hospitalization" will be defined as hospitalization for any non-surgical reason occurring within the last 3 months before assessment. The "stage" of cancer will be dichotomized into two categories: "local stage" and "advanced stage." The latter will be composed of "locally advanced and metastatic disease." The "time since cancer diagnosis" will refer to the time between the day of the assessment and the objective first diagnosis of the cancer or the recurrence of the cancer (if the patient was in complete remission). The "anti-hormonal therapy" will refer exclusively to the treatments recommended for women with hormone receptor positive breast cancer.

Clinical implications This study aims to evaluate the incidence and study the association between arterial thromboembolism and occult cancer. Moreover, this study will provide a RAM for arterial thrombosis applicable to cancer patients at any time after anticancer therapy initiation

ELIGIBILITY:
Inclusion Criteria:Ambulatory cancer patients, with histologically confirmed solid cancer (breast, lung, gastric, colorectal, pancreatic, ovarian, prostate, or bladder cancer) or specific hematologic malignancy (Hodgkin and non-Hodgkin lymphoma or multiple myeloma) -

Exclusion Criteria: a) age younger than 18 years, (b) life expectancy less than 3 months, (c) ongoing pregnancy, (d) recent (≤3 months) arterial thromboembolism and/or (e) major psychiatric disorder will be excluded from the study.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory cancer patients, with histologically confirmed solid cancer (breast, lung, gastric, colorectal, pancreatic, ovarian, prostate, or bladder cancer) or specific hematologic malignancy (Hodgkin and non-Hodgkin lymphoma or multiple myeloma). Patients diagnosed with multiple primary cancers during the study period will be assigned to the cancer type diagnosed first.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite of symptomatic arterial thromboembolism (any inpatient diagnosis) | 2 years
  a. acute coronary syndrome (ACS) including ST- elevation myocardial infarction (STEMI), non-ST elevation MI (NSTEMI) or unstable angina (UA), b. transient ischemic attack (TIA) or ischemic stroke or c. other arterial thromboembolism (systemic embolism or mesenteric ischemia) defined according to the respective diagnostic criteria and recommendations.

SECONDARY OUTCOMES:
Peripheral arterial disease | 2 years
  Diagnosis or progression peripheral artery disease
Hypertension | 2 years
  New or worsening hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Konstantinos Toutouzas, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Abdol Razak, N., Jones, G., Bhandari, M., Berndt, M. & Metharom, P. Cancer-Associated Thrombosis: An Overview of Mechanisms, Risk Factors, and Treatment. Cancers (Basel). 10, 380 (2018). 2. Blann, A. D. & Dunmore, S. Arterial and venous thrombosis in cancer patients. Cardiol. Res. Pract. 2011, 394740 (2011). 3. Di Nisio, M. et al. Arterial thrombosis in ambulatory cancer patients treated with chemotherapy. Thromb. Res. 127, 382-383 (2011). 4. Gerotziafas, G. T., Papageorgiou, L., Salta, S., Nikolopoulou, K. & Elalamy, I. Updated clinical models for VTE prediction in hospitalized medical patients. Thromb. Res. 164, S62-S69 (2018). 5. De Stefano, V. Arterial thrombosis and cancer: the neglected side of the coin of Trousseau syndrome. Haematologica 103, 1419-1421 (2018). 6. Aronson, D. & Brenner, B. Arterial thrombosis and cancer. Thromb. Res. 164, S23-S28 (2018). 7. Tuzovic, M. et al. Arterial Thrombosis in Patients with Cancer. Curr. Treat. Options Cardiovasc. Med. 20, 40 (2018). 8. Frere, C., Martin-Toutain, I., Thuny, F. & Bonello, L. Risk of Arterial Thrombosis in Cancer Patients. J. Am. Coll. Cardiol. 71, 260 (2018). 9. Hung, Y.-S. et al. Incidence, Risk Factors, and Outcomes of Arterial Thromboembolism in Patients with Pancreatic Cancer Following Palliative Chemotherapy. Cancers (Basel). 10, (2018). 10. Navi, B. B. et al. Risk of Arterial Thromboembolism in Patients With Cancer. J. Am. Coll. Cardiol. 70, 926-938 (2017). 11. Oren, O. & Herrmann, J. Arterial events in cancer patients-the case of acute coronary thrombosis. J. Thorac. Dis. 10, S4367 (2018). 12. Grilz, E. et al. Frequency, risk factors, and impact on mortality of arterial thromboembolism in patients with cancer. Haematologica 103, 1549-1556 (2018). 13. Baron, J. A., Gridley, G., Weiderpass, E., Nyren, O. & Linet, M. Venous thromboembolism and cancer. Lancet 351, 1077-1080 (1998). 14. Gregson, J. et al. Cardiovascular Risk Factors Associated With Venous Thromboembolism. JAMA Cardiol. 4, 163 (2019). 15. Abdel-Razeq, H. et al. Thromboembolic events in cancer patients on active treatment with cisplatin-based chemotherapy: another look! Thromb. J. 16, 2 (2018). 16. Gerotziafas, G. T. et al. A Predictive Score for Thrombosis Associated with Breast, Colorectal, Lung, or Ovarian Cancer: The Prospective COMPASS-Cancer-Associated Thrombosis Study. Oncologist 22, 1222-1231 (2017). 17. Antic, D. et al. Development and validation of multivariable predictive model for thromboembolic events in lymphoma patients. Am. J. Hematol. 91, 1014-1019 (2016). 18. Boura, P. et al. PO-53 - Prospective evaluation of risk assessment models and biological markers of hypercoagulability for the identification of high VTE risk patients with lung adenocarcinoma. The ROADMAP study. Thromb. Res. 140, S196 (2016). 19. Anand, L. N. et al. External validation of the COMPASS-Cancer Associated Thrombosis Study: A predictive score to identify patients with solid tumors on treatment who are at risk for venous thromboembolism. J. Clin. Oncol. 37, e18005-e18005 (2019). 20. WHO | International Classification of Diseases for Oncology, 3rd Edition (ICD-O-3). WHO (2019). 21. Austin, P. C. & Steyerberg, E. W. Events per variable (EPV) and the relative performance of different strategies for estimating the out-of-sample validity of logistic regression models. Stat. Methods Med. Res. 26, 796 (2017).